CLINICAL TRIAL: NCT00406523
Title: A Single Center Prospective Randomized Controlled Clinical Study of JANUS Stent in Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH-2006-B003
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Device: JANUS Stent

SUMMARY:
Janus stent is the only marketed drug-eluting stent (DES) without polymer coating as yet in China. The goal of this study is to evaluate the efficacy of JANUS (Tacrolimus eluted stent) in inhibiting of restenosis in percutaneous coronary intervention (PCI) real world and to observe the safety and efficacy of 4 months'clopidogrel treatment after implantation of JANUS stent.

Patients were enrolled and randomized to be treated by JANUS or SRNCRO (bare metal stent with the same platform as JANUS). All enrolled patients received daily clopidogrel for 4 months and aspirin for life long for post-PCI period(In AMI group, patients received daily clopidogrel 150mg for 2 weeks at first). The primary endpoints included death of heart, myocardial infarction, revascularization of the target lesson, sub-acute and late stent thrombosis one year after PCI, The secondary endpoints included MACE at 30 days, 6 months and restenosis by follow-up angiogram at 6 to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were eligible for coronary stenting
* All patients enrolled were implanted only one kind of stent
* Stent number ≤ 8 per patient and ≤3 per vessel (stents overlapping part for 3～5mm and being fully post-dilated; Total stent length ≤ 85mm in same vessel)
* Willing and able to sign informed consent.

Exclusion Criteria:

* Patients with multi-vessel disease could not be implanted the same kind of stent
* In-stent restenosis target lesion
* Patients not eligible for DES implantation (e.g. intolerance to anti-platelet therapy or undergoing heart or non-heart surgery recently

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-02; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, M.D., Principal Investigator — Shenyang Northern Hospital